CLINICAL TRIAL: NCT07299188
Title: The Effect of Using Electrically Insulated Gloves During Defibrillation on ROSC (Return of Spontaneous Circulation) Time, End-tidal CO₂ (EtCO₂) Response, Survival and Morbidity for Uninterrupted CPR: A Prospective Controlled Study in Manikins and Humans
Brief Title: Effect of Electrically Insulated Gloves on ROSC Time, End-tidal CO₂ Response, Survival and Morbidity in Uninterrupted CPR
Acronym: IG-CPR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ejder Saylav BORA, Assoc. Prof. M.D. PhD, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IzmirKCU-EM-01
Record Dates: First submitted 2025-11-24; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cardiopulmonary Resuscitation (CPR); Electrical Shock; Defibrillation
Keywords: Cardiopulmonary resuscitation; electrically insulated composite gloves; Uninterrupted resuscitation during defibrillation

STUDY DESIGN:
Intervention Model Description: EN 60903:2003 and IEC 60903:2014 compliant, Class 2 (17,000 V AC) electrically insulated composite Starline Linepro insulation gloves will be used. These gloves were chosen because they offer advantages to the rescuer in terms of high insulation capacity, flexible structure, and maneuverability during CPR. With the use of these gloves, the rescuer will be able to continue chest compressions without interruption during defibrillation, without breaking physical contact with the patient. This application will be evaluated in terms of both electrical safety and resuscitation quality.
  A total of 32 patients who have suffered cardiac arrest in the emergency department and whose initial rhythm is shockable (ventricular fibrillation or pulseless ventricular tachycardia) will be included in the study. Patients will be divided into two groups: an experimental group (n=16) receiving uninterrupted CPR protocol and a control group (n=16) receiving standard CPR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): GROUP WHICH LL BE APPLIED STANDARD CPR PROTOCOL OF AHA BUT WİTHOUT ELECTRİCALLY ISOLATED GLOVES
- INTERVENTION GROUP (Active Comparator): HAND ON DEFIBRILLATION GROUP (WITH GLOVES)
  Interventions: Device: HANDS ON BUT OFF DEFIBRILLATION

INTERVENTIONS:
Device: HANDS ON BUT OFF DEFIBRILLATION — GROUP WHICH LL BE APPLIED STANDARD CPR PROTOCOL OF AHA BY USING ELECTRICALLY ISOLATED GLOVES
  Arms: INTERVENTION GROUP

SUMMARY:
Cardiopulmonary arrest is the sudden cessation of spontaneous breathing and circulation due to various causes. Cardiopulmonary resuscitation (CPR) is the set of decisions and procedures encompassing all efforts aimed at restoring spontaneous circulation. Guidelines are published at regular intervals by the American Heart Association (AHA) and the European Resuscitation Council (ERC) to ensure that these procedures are applied uniformly worldwide. According to the AHA and ERC guidelines, the latest approach to CPR is to reduce the duration of interruptions in chest compressions, which is a component of high-quality CPR. Prior to actual patient intervention, a preliminary test will be conducted on an advanced life support simulation manikin to evaluate the safety and feasibility of the method.

During cardiopulmonary resuscitation (CPR), unavoidable interruptions in chest compressions occur because contact with the patient must be broken during defibrillation and cardioversion. In this study, electrically insulated composite gloves (Class 2) will be used to ensure uninterrupted chest compressions during defibrillation, and the effect of this practice on patients' ROSC, EtCO₂, neurological outcomes, and survival rates will be evaluated comparatively with the control group.

The main objective of the study is to evaluate the effect of ensuring uninterrupted chest compressions during defibrillation using electrically insulated composite gloves on patient survival rates.

DETAILED DESCRIPTION:
High-quality cardiopulmonary resuscitation (CPR) performed in cases of cardiac arrest is a determinant of survival and neurological outcomes. In this context, the quality and continuity of chest compressions are considered to be parameters that directly affect return of spontaneous circulation (ROSC) and long-term survival. Current guidelines strongly recommend that chest compressions be performed continuously and that compression intervals be kept to a minimum. This is because each pause causes a significant decrease in coronary and cerebral perfusion and prolongs the time required to restore effective circulation.

Although defibrillation during CPR is vitally important, especially in shockable rhythms, chest compressions are stopped during this procedure for the rescuer's safety, leading to a temporary interruption of circulation. The literature shows that compression interruptions before and after defibrillation reduce ROSC rates, lower end-tidal CO₂ (EtCO₂) levels, and have negative effects on overall survival. Therefore, the goal is to perform all interventions during CPR, including defibrillation, as quickly as possible and without interrupting chest compressions.

Before starting this study, a preliminary test was planned on a full-body simulation manikin used in advanced life support training to evaluate the safety of the method and materials to be used. The application of uninterrupted chest compressions during defibrillation using EN 60903 Class 2 insulated gloves will be tested on this manikin; the safety of the application, equipment durability, and feasibility from the rescuer's perspective will be observed. The findings obtained will provide a preliminary assessment of the method's suitability for field conditions before proceeding to work on patients.

Recent studies have shown that when gloves providing adequate electrical insulation are used, rescuers can safely continue chest compressions during defibrillation. It has been demonstrated that electrically insulated composite gloves with high insulation properties can effectively protect the rescuer by providing resistance to defibrillation voltages. However, standard medical examination gloves do not provide adequate protection against such high voltages; simulation studies have reported that many gloves fail at voltages between 2500-4000 V, posing a risk to rescuer safety. The voltage-current relationship of different types of gloves was evaluated, and it was shown that even double-layered latex gloves allowed current to pass through at a rate of 77% against external defibrillation voltage. These findings highlight the need to use not only insulated but also highly durable special gloves to ensure the safe application of defibrillation during CPR.

Although some third-level emergency departments and intensive care units now have automated CPR devices, access to these devices can be difficult nationwide. This study was designed based on the idea that the use of electrically resistant gloves to protect against electric shock during defibrillation after detectable rhythm detection for uninterrupted CPR would prevent interruption of perfusion, which is the main goal.

This study aims to evaluate the effects of maintaining uninterrupted chest compressions even during defibrillation during CPR on ROSC time, EtCO₂ levels, short- and long-term survival rates, and morbidity, based on the results of a 3-year study. The findings obtained may contribute to optimizing clinical practice by more clearly demonstrating the importance of uninterrupted CPR in advanced life support algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with in-hospital cardiac arrest requiring CPR
* Patients with shockable rhythms (pulseless ventricular tachycardia (VT) and ventricular fibrillation (VF))
* Adult patients aged 18 years and older
* Patients capable of providing informed consent or for whom consent can be obtained through a legal representative

Exclusion Criteria:

* Out-of-hospital cardiac arrests
* Patients who received CPR outside the emergency department
* Traumatic patients
* Pregnant patients
* Patients under 18 years of age
* Terminally ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-10-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
MORTALITY RATE | UP TO 36 MONTHS
  The study will be conducted using electrically insulated composite gloves (Class 2 Starline Linepro insulated gloves) to ensure that chest compressions continue uninterrupted during defibrillation and to determine the effect of this practice on patient survival rates.

SECONDARY OUTCOMES:
ROSC (return of spontaneous circulation) times | UP TO 36 MONTHS
  At what time interval could ROSC be achieved with non-conductive gloves during CPR compared to the control group?
End-tidal carbon dioxide (EtCO₂) response | UP TO 36 MONTHS
  EtCO₂ levels during CPR with or without insulated gloves (mmHg)
Its effect on post-CPR neurological outcomes will be evaluated | UP TO 36 MONTHS
  post-CPR neurological outcomes with or without insulated gloves (modified ranking score (0-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang T, Sun Y, Zhang H, Zhang Q, Tang S, Niu X, Guo Y, Li K, Chen Y, Xu F. Combined end-tidal CO2 and diastolic blood pressure-guided CPR improves survival from cardiac arrest in porcine model. Resuscitation. 2025 Nov;216:110745. doi: 10.1016/j.resuscitation.2025.110745. Epub 2025 Aug 5. PMID 40752672
- [Background] Deakin CD, Lee-Shrewsbury V, Hogg K, Petley GW. Do clinical examination gloves provide adequate electrical insulation for safe hands-on defibrillation? I: Resistive properties of nitrile gloves. Resuscitation. 2013 Jul;84(7):895-9. doi: 10.1016/j.resuscitation.2013.03.011. Epub 2013 Mar 16. PMID 23507464
- [Background] Musiari M, Saporito A, Ceruti S, Biggiogero M, Iattoni M, Glotta A, Cantini L, Capdevila X, Cassina T. Can a Glove-Coach Technology Significantly Increase the Efficacy of Cardiopulmonary Resuscitation on Non-healthcare Professionals? A Controlled Trial. Front Cardiovasc Med. 2021 Dec 9;8:685988. doi: 10.3389/fcvm.2021.685988. eCollection 2021. PMID 34957226
- [Background] Deakin CD, Thomsen JE, Lofgren B, Petley GW. Achieving safe hands-on defibrillation using electrical safety gloves--a clinical evaluation. Resuscitation. 2015 May;90:163-7. doi: 10.1016/j.resuscitation.2014.12.028. Epub 2015 Feb 26. PMID 25725295